CLINICAL TRIAL: NCT07254143
Title: Clinical And Radiographic Efficacy Of MTA Flow In Apicoectomy
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: 175 Military hospital (Unknown)
Responsible Party: Principal Investigator, Son Hoang Le, Lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 493/HĐĐĐ-ĐHYD
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Clinical and Radiographic Success in 6 Months
Keywords: Apicoectomy; Retrograde filling; MTA Flow™; Mineral trioxide aggregate; Periapical healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- MTA flow: MTA flow group have this material for retrograde filling in apicoectomy.
  Interventions: Drug: MTA flow material

INTERVENTIONS:
Drug: MTA flow material — This group is used MTA flow material for retrograde filling in apicoectomy.

SUMMARY:
The goal of this observational study is to learn about the short-term effects of MTA flow thick material in apicoectomy treatment. Participants are patients who take MTA flow to treat their apical lesion. The main question it aims to answer is:

Is MTA flow thick material effective for retrograde filling in patients who require apicoectomy for treating apical lesion? Participants already taking MTA flow as part of their regular dental care for apicoectomy will be followed-up treatment results in 6 months.

DETAILED DESCRIPTION:
Quality assurance plan: all patients satisfy the inclusion criteria are invinted to participate the study. Radiography was performed using an standard kit. All surgical procedures were conducted by an experienced oral surgeon. Clinical signs, radiographic signs are independently evaluated by an endodontist and oral surgeon.

Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification: medical records adn paper report form. Data dictionary: clinical signs, swelling, pain, fistula, radiographic signs, success rate, rarefaction, periodontal space.

Standard Operating Procedures: none. Sample size assessment: none available. Plan for missing data: exclude from the participants, missing case will be reported in the results.

Statistical analysis plan: Data were collected and analysed using JASP software, version 0.19.3 (University of Amsterdam, Amsterdam, The Netherlands). Categorical variables are presented as absolute counts and percentages, whereas numerical variables are expressed as mean values with standard errors.

The Friedman test was used to compare differences in clinical symptoms and apical lesion sizes at baseline, 3 months, and 6 months. The Bonferroni post hoc test was used for pairwise comparisons between assessment points. The chi-square test was used to compare the differences in radiographic findings and overall success between 3-month and 6-month evaluations.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* systemic health classified as I or II according to the American Society of Anesthesiologists (ASA) classification
* willingness to participate in the study
* failure of conventional or repeat endodontic treatment
* a periapical lesion with a diameter ≥ 5 mm

Exclusion Criteria:

* a crown-to-root ratio ≥ 1.0
* inability to comply with the follow-up protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population are patients who came to Dental Department of 175 Military hospital for apical lesions.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical success | 6 months
  Clinical success is defined as absence of 4 clinical signs. These clinical signs included pain, swelling, and fistula at the etiologic tooth.
Radiographic success | 6 months
  To evaluate healing progression on periapical radiographs, images obtained at 3 and 6 months were compared with those taken at 7 days post-surgery. Radiographic success was evaluated according to the criteria proposed by Rud et al. (1972) and Molven et al. (1987).

CONTACTS AND LOCATIONS:
Overall Officials: Loan-Chi Thi Bui, Principal Investigator — Military Hospital 175
Locations (1):
- Military Hospital 175, Hanh Thong Ward, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared when other researchers ask for specific purpose.